CLINICAL TRIAL: NCT01037023
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance (PMS) to Monitor the Safety and Effectiveness of HYCAMTIN Administered in Korean Patients According to the Prescribing Information
Brief Title: Regulatory Hycamtin(Oral) PMS
Acronym: Hycamtin PMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113946
Record Dates: First submitted 2009-12-10; First posted 2009-12-21 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Lung Cancer, Small Cell
Keywords: PMS (post-marketing surveillance); Topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients administrated Topotecan: There is only one group. This group includes patients administrated Topotecan
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Topotecan — patients administrated Topotecan according to the prescribing information

SUMMARY:
Non-interventional, open-label, single group, multicentric post-marketing surveillance to monitor the safety and effectiveness of Topotecan administered in Korean patients according to the prescribing information

DETAILED DESCRIPTION:
Non-interventional, open-label, single group, multicentric post-marketing surveillance to monitor the safety and effectiveness of Topotecan administered in Korean patients according to the prescribing information

Topotecan will be administered as described the prescribing information or by physician's decision.

ELIGIBILITY:
All subjects must satisfy the following criteria.

* Subject who is under the indication to the prescribing information of oral Hycamtin.
* Subject who is treated with oral Hycamtin according to the judgement of her or his investigator.

All subjects must not satisfy the following criteria.

• Subject who is under the contraindication to the prescribing information of oral Hycamtin.

As considering the characteristic of observational post marketing surveillance, the exclusion criteria is not strict. All investigators should prescribe oral Hycamtin according to prescribing information which approved in Korea.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients administrated Topotecan at the site
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2010-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events after Topotecan administration | 9 months

SECONDARY OUTCOMES:
Occurrence of unexpected adverse event or adverse drug reaction | 9 months
Occurrence of serious adverse event or adverse drug reation | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- South Korea (2):
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul